CLINICAL TRIAL: NCT01064609
Title: "Diagnostic Yield and Safety of Transbronchial Lung Biopsy Using Cryoprobes Versus Conventional Forceps:a Randomized Clinical Trial"
Brief Title: "Diagnostic Yield and Safety of Transbronchial Lung Biopsy Using Cryoprobes Versus Conventional Forceps.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-003232-38
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2011-06

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2. Biopsy with cryoprobes (Active Comparator): Transbronchial cryobiopsy with a cryoprobe.
  Interventions: Procedure: Biopsy by cryoprobes
- 2.Biopsy with forceps (Active Comparator): Transbronchial lung biopsy with conventional forceps.
  Interventions: Procedure: Biopsy with conventional forceps

INTERVENTIONS:
Procedure: Biopsy by cryoprobes — Transbronchial lung biopsy with cryoprobes.
  Arms: 2. Biopsy with cryoprobes
Procedure: Biopsy with conventional forceps — Transbronchial lung biopsy with conventional forceps.
  Arms: 2.Biopsy with forceps

SUMMARY:
Transbronchial lung biopsy (TBLB) is a bronchoscopic procedure used to obtain peripheral lung tissue. Small size and artefacts cause variable, and usually poor, diagnostic yield. The use of cryoprobes may allow for larger size and better quality biopsy samples.

Objectives:To analyze the histological quality and immunohistochemical findings of samples obtained by cryoprobe compared with TBLB obtained by conventional forceps and to assess the safety and complications of TBLB with cryoprobe versus the conventional method.

Methodology:

Prospective randomized study of 80 patients. The transbronchial lung biopsy was indicated for diagnoses of a interstitial lung disease. In both procedures the videobroncoscopy used will be a Olympus 260-T.

The transbronchial lung biopsy will be carried out with conventional forceps (Boston ® Biopsy Forceps, Ref 1556 and Olympus ® FB-19E) and cryoprobe (Erbokryo AC ®). TBLB will be performed by fluoroscopy guided and the cryoprobe or forceps will place in an area of the peripheral lung previously selected according to CT findings. Lung biopsies will be processed: The samples submitted for histological analysis will be fixed in formalin and embedded in paraffin. Staining will perform with hematoxylin-eosin and Masson's trichrome and the samples will be analyzed by a pathologist according to a protocol. The samples submitted to immunohistochemical study will be frozen (liquid nitrogen) for later transport.The specifical monoclonal antibodies will be used for immunohistochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Interstitial Lung disease.

Exclusion Criteria:

* Respiratory failure,haemodynamic instability, haemoptysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To analyze the histological quality and immunohistochemical findings of samples obtained by cryoprobe compared with TBLB obtained by conventional forceps. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pajares, Doctor, Principal Investigator — Hospital del Santa Creu i Sant Pau; Alfons Torrego, Doctor, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Mª Carmen Puzo, Doctor, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Sanrta Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Pajares V, Puzo C, Castillo D, Lerma E, Montero MA, Ramos-Barbon D, Amor-Carro O, Gil de Bernabe A, Franquet T, Plaza V, Hetzel J, Sanchis J, Torrego A. Diagnostic yield of transbronchial cryobiopsy in interstitial lung disease: a randomized trial. Respirology. 2014 Aug;19(6):900-6. doi: 10.1111/resp.12322. Epub 2014 Jun 1. PMID 24890124